CLINICAL TRIAL: NCT05784922
Title: Health Opportunities and Promoters of Equitable Screening for Lung Cancer (HOPES for Lung Cancer)
Brief Title: Health Opportunities and Promoters of Equitable Screening for Lung Cancer
Acronym: HOPES
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Efren J. Flores, M.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 1K08CA270430-01A1 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer; Smoking Behaviors; Diagnosis
Keywords: lung cancer screening; Hispanic outreach; educational intervention; digital health; smoking documentation; smoking history; health equity
MeSH Terms: conditions — Lung Neoplasms; Smoking; Disease | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Digital Outreach: Patient Gateway: Participants who list "Patient Gateway" as the preferred mode of contact in the electronic health record (EHR) system. Patient Gateway is an online patient portal that gives patients access to securely message their Mass General Brigham provider, request routine appointments, prescriptions and referral authorizations as well as view test results that were processed at a Mass General Brigham facility. Participants will receive the digital educational lung cancer screening video via their patient gateway account.
  Interventions: Other: Educational Lung Cancer Screening (LCS) Video
- Digital Outreach: Text: Participants who list "Text" as the preferred mode of contact in the electronic health record (EHR) system. Participants will receive the digital educational lung cancer screening video via a text message sent directly to their cell phone.
  Interventions: Other: Educational Lung Cancer Screening (LCS) Video
- Digital Outreach: Email: Participants who list "Email" as the preferred mode of contact in the electronic health record (EHR) system. Participants will receive the digital educational lung cancer screening video directly to the email they have listed.
  Interventions: Other: Educational Lung Cancer Screening (LCS) Video

INTERVENTIONS:
Other: Educational Lung Cancer Screening (LCS) Video — An educational video on lung cancer screening tailored to Hispanic current and former smokers.

SUMMARY:
The goal of this clinical trial is to promote lung cancer screening (LCS) uptake among Hispanic current and former smokers. The main questions it aims to answer are:

* What barriers do current and former Hispanic smokers face in the identification and documentation of their smoking status?
* How can digital delivery of an educational video promote LCS uptake among current and former Hispanic smokers?

Participants will receive an educational video about lung cancer screening and complete brief, self-reported surveys afterwards.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-specific mortality in the US, and Hispanics experience worse lung cancer outcomes and die at higher rates due to advanced stage at presentation. Lung cancer screening (LCS) can save many lives through early lung cancer detection among Hispanic current and former smokers.

Still, without increasing efforts to improve smoking status disclosure and documentation and tailored interventions to promote LCS uptake among Hispanic current and former smokers, this underserved population will continue to demonstrate disparities in lung cancer survival. Based on prior research experience, Dr. Flores has adapted the NIMHD research framework by incorporating elements from Ford's evidence-based theoretical model to guide the following proposed study aims:

1) To elucidate barriers and facilitators to consistent identification and documentation of smoking status to promote LCS uptake among Hispanic current and former smokers; 2) To assess feasibility, acceptability, and reach of the digital delivery of an educational video to promote LCS uptake among Hispanic current and former smokers; 3) To explore the effect of the digital delivery of the educational video to increase interest, intent, and scheduling of LCS uptake among Hispanic current and former smokers.

Impact: The successful completion of this research will serve as a foundation for developing novel interventions to overcome disparities and advance equity in lung cancer outcomes among Hispanics and other vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Must be 50-80 years old
* Are a current or former smoker (quit within 15 years, or a cumulative smoking status of > 20 pack-years)
* Not currently enrolled in Lung Cancer Screening
* Must speak English or Spanish

Exclusion Criteria:

* Has a clinical cognitive inability to provide informed consent for participation in the study or complete a brief survey
* Currently diagnosed with lung cancer
* Currently enrolled in lung cancer screening
* Have participated in the focus groups discussions from Aim 1

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators chose to restrict eligibility to adults aged 50-80 with no personal history of lung cancer to meet the United States Preventive Services Task Force Guidelines for lung cancer screening. As the primary aim of this study is to address the disparities in lung cancer screening rates and outcomes for Hispanic individuals, only Hispanic-identifying patients will be eligible for participation. Further grants stemming from this project will include community-based outreach efforts to extend the testing and dissemination of this intervention to other underrepresented groups.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Participant outreach (contact) of digital link | Year 3
  Reach is defined as >20% of enrolled participants interacting with the digital delivery of the LCS educational video (i.e., partial or complete review of the LCS educational video).

SECONDARY OUTCOMES:
Participant interaction with digital link | Year 3
  Overall proportion of participants that click on the embedded link to the successfully digitally delivered LCS educational videos
Participant attention of LCS video | Year 3
  Duration of viewing the LCS video (i.e., partial or complete)
Survey completion | Year 4
  Overall proportion of survey completion by participants.

OTHER OUTCOMES:
Participant baseline smoking status | Year 5
  Identify salient participant characteristics obtained from the EHR (e.g., smoking status) among those that interacted with the digital delivery modality.
Participant acceptability of intervention | Year 5
  Investigate attributes of the intervention to guide future research and development to create such an intervention (for future trials)

CONTACTS AND LOCATIONS:
Overall Officials: Efren Flores, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Narayan AK, Chowdhry DN, Fintelmann FJ, Little BP, Shepard JO, Flores EJ. Racial and Ethnic Disparities in Lung Cancer Screening Eligibility. Radiology. 2021 Dec;301(3):712-720. doi: 10.1148/radiol.2021204691. Epub 2021 Sep 21. PMID 34546133
- [Background] Percac-Lima S, Ashburner JM, Atlas SJ, Rigotti NA, Flores EJ, Kuchukhidze S, Park ER. Barriers to and Interest in Lung Cancer Screening Among Latino and Non-Latino Current and Former Smokers. J Immigr Minor Health. 2019 Dec;21(6):1313-1324. doi: 10.1007/s10903-019-00860-2. PMID 30701427
- [Background] Wang GX, Neil JM, Fintelmann FJ, Little BP, Narayan AK, Flores EJ. Guideline-Discordant Lung Cancer Screening: Emerging Demand and Provided Indications. J Am Coll Radiol. 2021 Mar;18(3 Pt A):395-405. doi: 10.1016/j.jacr.2020.08.005. Epub 2020 Sep 6. PMID 32905787
- [Background] Flores EJ, Park ER, Irwin KE. Improving Lung Cancer Screening Access for Individuals With Serious Mental Illness. J Am Coll Radiol. 2019 Apr;16(4 Pt B):596-600. doi: 10.1016/j.jacr.2018.12.045. PMID 30947893
- [Background] Irwin KE, Steffens EB, Yoon Y, Flores EJ, Knight HP, Pirl WF, Freudenreich O, Henderson DC, Park ER. Lung Cancer Screening Eligibility, Risk Perceptions, and Clinician Delivery of Tobacco Cessation Among Patients With Schizophrenia. Psychiatr Serv. 2019 Oct 1;70(10):927-934. doi: 10.1176/appi.ps.201900044. Epub 2019 Jul 30. PMID 31357921

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT05784922/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT05784922/ICF_001.pdf